CLINICAL TRIAL: NCT04931303
Title: Digital GaitCare - Therapy Monitoring in the Home Environment of Patients With Parkinson Via Digital Gait Analysis and Patient Feedback
Brief Title: Digital GaitCare - Therapy Monitoring in the Home Environment of Patients With Parkinson
Status: Completed | Type: Observational
Sponsor: Medical Valley Digital Health Application Center GmbH (Industry)
Collaborators: University Hospital Erlangen (Other); University of Regensburg (Other); Philipps University Marburg (Other); Hospital Rummelsberg (Unknown); NeuroPoint GmbH (Unknown); Portabiles HealthCare Technologies GmbH (Unknown); Systemhaus Ulm GmbH (Unknown); Fraunhofer Institute for Integrated Circuits IIS (Unknown); Friedrich-Alexander-Universität Erlangen-Nürnberg (Other); University of Luxembourg (Other); Leibniz Centre for European Economic Research GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2021-06-01; First posted 2021-06-18 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2021-06

CONDITIONS: Parkinson Disease; Gait Disorders, Neurologic
Keywords: Parkinson; Gait Analysis; Digital Health; Home-Monitoring
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Enrolled patients receive a medical device which monitors gait quality and collects information about the patients health status. Possible changes of intervention (drug or physical therapy) within the observational phase (8 weeks) are initiated and prescribed by physicians as a result of routine care process or patient contact based on their (deteriorated) health status. With the chosen endpoints, changes of patients empowerment, gait quality and system usability by using a monitoring device are monitored.

SUMMARY:
Gait disturbances and movement restrictions occur frequently in Parkinson's disease. Patient-centered monitoring with objective aids in the patient's daily life, supports and promotes therapy decisions made by physicians and patients. Technical, sensor-based monitoring has the potential to generate objective target parameters at any point in time during therapy (patient journey), representing the state of health and its progression, and to make this information available to physicians and patients via telemedical data management. In this study, the gait analysis system "Mobile GaitLab Home 2.0", consisting of sensors for gait data acquisition, a smartphone application for study participants (Mobile GaitLab app) and a web portal for physicians (Mobile GaitLab portal) is used for data collection.

The research question is divided into three sub-objectives: First, the study explores and tests how technically generated parameters of sensor-based gait analysis can map the symptom "bradykinesis". The second goal is the explorative investigation of how a tele-health service support with low-threshold access to medical professionals, can be integrated into the care process. The third goal is the implementation evaluation of the technological developments. Here, it is examined to determine the extent to which the implementation of gait data and patient feedback (PROMs) in the patient-centered care process within the framework of clinical decision support contributes to early gait-associated therapy optimization and thus improves the general health of patients and how initial indications of positive care effects for patients can be derived.

During a 60-day observation phase, study participants use the gait analysis system, which records their gait pattern throughout the day and collects data via the Mobile GaitLab app. Study participants are asked to perform standardized gait tests in the home environment several times a day, in addition to continuous measurements during the awake phase. Frequency of data collection is controlled by Mobile GaitLab Home 2.0 and can be flexibly adjusted to the study participant's health status and therapy. The Mobile GaitLab app uses questionnaires to record data on gait safety, activity, general well-being, and events relevant to the disease. An evaluation of these data (PROMs) and the results from the gait analyses, are visualized for the study participants via the Mobile GaitLab app.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease (H&Y I-IV)
* Age > 18 years
* Ability to walk > 4 x 10 m without assistance
* Ability to speak and read
* Ability to use an application that can be mapped on a smart device
* Informed consent of the study participant
* Willingness of the study participant to take therapy measures (e.g., medication therapy, exercise therapy)

Exclusion Criteria:

* Tremor-dominant Parkinson's syndrome without involvement of the lower extremities
* Aphasia and alexia
* Visual disturbances that make reading impossible
* Higher-grade movement disorders, with high risk of falls and non-independent ability to walk
* Higher grade cognitive deficits
* Inability of the study participant to understand the information and procedures of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be enrolled during their routine outpatient or physician visit or inpatient stay.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Difference in gait parameters (stride length) during 4x10 meter gait test (4x10m) performed at clinic | day 1 and day 60
  Difference in stride length in cm during 4x10m performed at clinic
Difference in gait parameters (stride time) during 4x10 meter gait test (4x10m) performed at clinic | day 1 and day 60
  Difference in stride time in seconds during 4x10m performed at clinic
Difference in gait parameters (gait speed) during 4x10 meter gait test (4x10m) performed at clinic | day 1 and day 60
  Difference in gait speed in m/s during 4x10m performed at clinic
Difference in gait parameters (heel-strike angle) during 4x10 meter gait test (4x10m) performed at clinic | day 1 and day 60
  Difference in heel-strike angle in degree during 4x10m performed at clinic
Difference in gait parameters (toe-off angle) during 4x10 meter gait test (4x10m) performed at clinic | day 1 and day 60
  Difference in toe-off angle in degree during 4x10m performed at clinic
Difference in gait parameters (foot-clearance) during 4x10 meter gait test (4x10m) performed at clinic | day 1 and day 60
  Difference in foot clearance in cm during 4x10m performed at clinic
Difference in gait parameters (variability) during 4x10 meter gait test (4x10m) performed at clinic | day 1 and day 60
  Difference in variability in percent during 4x10m performed at clinic
Difference in time of 1 x 10 meter gait test (1x10m) performed at baseline versus closeout | day 1 and day 60
  Difference in time, measured in seconds of 6 meter constant walking within the 10-meter gait test at baseline and at closeout
Difference in time of Timed-Up-and-Go Test (TUG) performed at baseline versus closeout | day 1 and day 60
  Difference in time, measured in seconds of TUG at baseline and at closeout
Difference in Unified Parkinson's Disease Rating Scale III (UPDRS III) Motor Score evaluated at baseline versus closeout | day 1 and day 60
  Difference in UPDRS III Motor Score (range from 0 to 56, Lower scores mean a better outcome) at baseline and at closeout
Difference in Shared-Decision-Making-Questionaire-9 (SDM-Q9) evaluated at baseline versus closeout | day 1 and day 60
  Difference in SDM-Q9 (range from 0 to 45, Higher scores mean a better outcome) at baseline and at closeout
Difference in Parkinsons-Disease-Questionaire (PDQ-39) evaluated at baseline versus closeout | day 1 and day 60
  Difference in PDQ-39 (range from 0 to 100, Lower scores mean a better outcome) at baseline and at closeout
Difference in Parkinson-specific-health-literacy evaluated at baseline versus closeout | day 1 and day 60
  Difference in Parkinson-specific-health-literacy (range from 0 to 100, Higher scores mean a better outcome) at baseline and at closeout
Number of useful Patient-Physician-Contacts evaluated at closeout | day 60
  Counted number of useful Patient-Physician-Contacts during study duration (range from 0 to individual number of Patient-Physician-Contacts) evaluated at closeout
System Usability Scale (SUS) and modified SUS evaluated at closeout | day 60
  SUS score per patient - range from 0 to 100 score points (Higher scores mean a better outcome.)
Collecting gait parameters (stride length) during gait tests and monitoring at home | day 1 to day 60
  Collection of gait parameters (stride length in cm)
Collecting gait parameters (stride time) during gait tests and monitoring at home | day 1 to day 60
  Collection of gait parameters (stride time in seconds)
Collecting gait parameters (gait speed) during gait tests and monitoring at home | day 1 to day 60
  Collection of gait parameters (gait speed in m/s)
Collecting gait parameters (heel-strike angle) during gait tests and monitoring at home | day 1 to day 60
  Collection of gait parameters (heel-strike angle in degree)
Collecting gait parameters (toe-off angle) during gait tests and monitoring at home | day 1 to day 60
  Collection of gait parameters (toe-off angle in degree)
Collecting gait parameters (foot clearance) during gait tests and monitoring at home | day 1 to day 60
  Collection of gait parameters (foot clearance in cm)
Collecting gait parameters (variability) during gait tests and monitoring at home | day 1 to day 60
  Collection of gait parameters (variability in percent)

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Winkler, Professor, Principal Investigator — Molekulare Neurologie, Universitätsklinikum Erlangen
Locations (5):
- Germany (5):
  - University Hospital Erlangen, Erlangen
  - Philipps University Marburg Medical Center, Marburg
  - University of Regensburg, Regensburg
  - Hospital Rummelsberg, Schwarzenbruck
  - Neuropoint GmbH, Ulm

IPD SHARING:
Plan to Share IPD: No